CLINICAL TRIAL: NCT03975387
Title: Phase 1/2 Open-Label Study of the Safety, Pharmacokinetics, and Preliminary Activity of ASTX295 in Subjects With Wild-Type TP53 Advanced Solid Tumors
Brief Title: Study of ASTX295 in Patients With Solid Tumors With Wild-Type p53
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTX295-01; 2021-005033-16 (EudraCT Number)
Record Dates: First submitted 2019-05-28; First posted 2019-06-05 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor
Keywords: solid tumor; mesothelioma; TP53
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASTX295 (Experimental)
  Interventions: Drug: ASTX295

INTERVENTIONS:
Drug: ASTX295 — ASTX295 orally for 28-day cycle continuous or on an intermittent dosing schedule.

SUMMARY:
Study ASTX295-01 is a first in human Phase 1/2 open-label study of the safety, pharmacokinetics, and preliminary activity of ASTX295 in participants with wild-type TP53 advanced solid tumors. Phase 1 is a dose escalation and dose expansion study design. Sponsor made the strategic decision to not pursue the Phase 2 part of the study.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be 18 years of age or older, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Have histologically or cytologically confirmed advanced solid tumors that are metastatic or unresectable and are refractory or have relapsed after treatment with standard available therapies or for whom standard life-prolonging measures are not available.

   1. Phase 1: any tumor type is eligible
   2. Phase 2: eligible tumor types as follows: malignant pleural mesothelioma (MPM) (Cohort 1); Liposarcoma (well-differentiated (WD) , de- differentiated (DD), or mix), intimal sarcoma, and other sarcomas with human murine double minute 2 (MDM2) amplification (Cohort 2); Glioblastoma multiforme (GBM) and tumors with CDNK2A loss of function (LOF) excluding MPM, liposarcoma, intimal sarcoma, and uveal melanoma (UVM) (Cohort 3); any solid tumors with molecular feature that may confer sensitivity to ASTX295 (Cohort 4); Uveal melanoma (Cohort 5); Any cancer type with MDM2 amplification excluding MPM, sarcoma, and UVM(Cohort 6).
3. Documented wild-type TP53 and other molecular feature requirements.
4. Have an Eastern Cooperative Oncology Group (ECOG) Performance status (PS) of 0 to 2.
5. Acceptable bone marrow function, as evidenced by the following laboratory data:

   1. Absolute neutrophil count (ANC) ≥1500 cells/mm3
   2. Platelet count ≥100,000 cells/mm3
   3. Hemoglobin >9 g/dL
6. Adequate hepatic function as evidenced by:

   1. Serum total bilirubin ≤1.5 × upper limit of normal (ULN).
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (≤ 3 ULN in the presence of liver metastases).
   3. Serum creatinine ≤1.5 × ULN OR calculated creatinine clearance (by the standard Cockcroft-Gault formula) of ≥50 mL/min or measured glomerular filtration rate of ≥50 mL/min.

   Sex
7. Participant can be male or female

   Informed Consent
8. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, and willing to participate in the study.

   Participants are eligible to be included in Phase 1 Part B of the study only if all of the following additional criteria apply:
9. In Phase 1 Part B (dose expansion) of the protocol, subjects must have disease lesions that are amenable to biopsy and must agree and be able to undergo a pre- and on- treatment biopsy.

   Participants are eligible to be included in Phase 2 of the study only if all of the following additional criteria apply:
10. Have sufficient tumor specimen either from archival formalin-fixed, paraffin embedded (FFPE) tissue or tissue obtained by a fresh biopsy for analyzing TP53 at a central laboratory.
11. Measurable disease according to appropriate criteria as per protocol.

Exclusion Criteria:

Medical Conditions

1. Poor medical risk in the investigator's opinion because of systemic diseases in addition to the cancer under study, for example, uncontrolled infections.
2. Life-threatening illness, significant organ system dysfunction, or other condition that, in the investigator's opinion, could compromise subject safety, or the integrity of study outcomes, or interfere with the absorption or metabolism of ASTX295.
3. History of, or at risk for, cardiac disease, as evidenced by any of the following conditions:

   1. Abnormal left ventricular ejection fraction.
   2. Congestive cardiac failure of ≥Grade 3.
   3. Unstable cardiac disease.
   4. History or evidence at Screening of long QT interval corrected for heart rate (QTcF), ventricular arrhythmias, clinically significant bradyarrhythmias, third-degree atrioventricular (AV) block, presence of cardiac pacemaker or defibrillator, or other clinically significant arrhythmias.
   5. Screening 12-lead electrocardiogram (ECG) with measurable QTcF interval of ≥470 msec. (Fridericia's formula should be used).
4. Known advanced human immunodeficiency virus (HIV) infection (including AIDS): clinical stage ≥ 3 according to WHO classification and/or HIV-associated immunodeficiency.
5. Known active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection (Inactive Hepatitis Carrier and subjects with laboratory evidence of no active replication on antivirals - viral load below limit of detection- will be permitted).
6. Known brain metastases, unless previously treated and clinically stable for at least 4 weeks with or without steroids.
7. Known significant mental illness or other conditions, such as active alcohol or other substance abuse that, in the opinion of the investigator, predispose the subject to high risk of noncompliance with the protocol treatment or assessments.

   Prior/Concomitant Therapy
8. Prior anticancer treatments or therapies within the indicated time window prior to first dose of study treatment (ASTX295), as follows:

   1. Cytotoxic chemotherapy within 3 weeks prior. Any encountered treatment-related toxicities (excepting alopecia) must be stabilized or resolved to ≤Grade 1.
   2. Monoclonal antibodies, biologics, or immunotherapy within 4 weeks prior. Any encountered treatment-related toxicities must be stabilized or resolved to ≤Grade 1.
   3. Molecularly targeted drug or other investigational drugs, without the potential for delayed toxicity, within 4 weeks of the first dose of study treatment or 5 half-lives (minimum 14 days), whichever is shorter. Any encountered treatment-related toxicities must be stabilized or resolved to ≤Grade 1.
   4. Major surgery or radiation within 4 weeks prior to first dose (palliative radiotherapy to a single lesion within 2 weeks).
9. Prior treatment with MDM2 antagonist
10. Inability to swallow oral medication or inability or unwillingness to comply with the administration requirements related to ASTX295.

    Participants are excluded from the Phase 2 part of the study if any of the following additional criteria apply:
11. Active malignancy other than the cancer under study (excludes low risk prostate cancer or early breast cancer with or without hormonal therapy, basal cell carcinoma of the skin and superficial bladder cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Safety and tolerability of ASTX295 including determination of maximum tolerated dose (MTD), and/or recommended dose for expansion (RDE) to Phase 1b | From the date of the first dose until 30 days after discontinuation of study treatment
Phase 1b: Recommended Phase 2 dose (RP2D) and regimen of ASTX295 to proceed to Phase 2 | From the date of the first dose until 30 days after discontinuation of study treatment, an average of 6 months to 1 year
  The RP2D will be based on incidence and severity of AEs, including SAEs and will be determined by the data and safety review committee (DSRC)
Phase 2: Disease control rate (DCR) in Cohort 1 | From the date of the first dose until Week 16
  DCR will be calculated in Cohort 1 as the number of subjects whose response at Week 16 is CR, partial response (PR), or stable disease, divided by the total number of subjects evaluable for DCR analysis.
Phase 2: Overall response rate (ORR) in Cohorts 2, 3, 4, 5, and 6 | From the date of the first dose until study treatment discontinuation, an average of 6 months to 1 year
  ORR in Cohorts 2, 3, 4, 5, and 6 will be calculated as the number of subjects whose best response is CR or PR, divided by the total number of subjects evaluable for ORR analysis.

SECONDARY OUTCOMES:
Phase 1: Preliminary clinical activity of ASTX295 as assessed by disease control rate (DCR) | From the date of the first dose until Week 16
  DCR will be calculated as the number of subjects whose response at Week 16 is CR, PR, or stable disease, divided by the total number of subjects evaluable for DCR analysis
Phase 1: Preliminary clinical activity as assessed by objective response rate (ORR) of ASTX295 | From the date of the first dose until study treatment discontinuation, an average of 6 months to 1 year
  ORR will be calculated as the number of subjects whose best response is CR or PR, divided by the total number of subjects evaluable for ORR analysis
Phase 2: Safety profile of ASTX295 | From the date of the first dose until 30 days after discontinuation of study treatment, an average of 6 months to 1 year
  Incidence and severity of adverse events (AEs) including serious adverse events (SAEs)
Phase 2: Progression free survival (PFS) | Up to approximately 1 year
  PFS is defined as the time from date of the first dose until the earliest date of disease progression or death from any cause, whichever comes first
Phase 2: Overall survival (OS) | Up to approximately 1 year
  OS is defined as the time from the date of first dose to date of death due to any cause
Phase 2: Overall response rate (ORR) in Cohort 1 | From the date of the first dose until study treatment discontinuation, an average of 6 months to 1 year
  ORR in Cohort 1 will be calculated as the number of subjects whose best response is CR or PR, divided by the total number of subjects evaluable for ORR analysis.
Pharmacokinetic (PK) profile of ASTX295 (area under the curve [AUC]) | Blood will be collected during Cycles 1 and 2 in Phase 1, Cycles 1 and 3 in Phase 2 (each cycle is 28 days)
Pharmacokinetic (PK) profile of ASTX295 (minimum concentration [Cmin]) | Blood will be collected during Cycles 1 and 2 in Phase 1, Cycles 1 and 3 in Phase 2 (each cycle is 28 days)
Pharmacokinetic (PK) profile of ASTX295 (maximum concentration [Cmax]) | Blood will be collected during Cycles 1 and 2 in Phase 1, Cycles 1 and 3 in Phase 2 (each cycle is 28 days)
Pharmacokinetic (PK) profile of ASTX295 (time to reach maximum concentration [Tmax]) | Blood will be collected during Cycles 1 and 2 in Phase 1, Cycles 1 and 3 in Phase 2 (each cycle is 28 days)
Pharmacokinetic (PK) profile of ASTX295 (elimination half-life [t½]) | Blood will be collected during Cycles 1 and 2 in Phase 1, Cycles 1 and 3 in Phase 2 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - City of Hope Comprehensive Cancer Center Site#114, Duarte, California
  - Cedars-Sinai Medical Center Site #105, Los Angeles, California
  - Hoag Hospital Site#110, Newport Beach, California
  - Holden Comprehensive Cancer Center Site#108, Iowa City, Iowa
  - University of Michigan Rogel Cancer Center Site#109, Ann Arbor, Michigan
  - Regions Cancer Center Site #115, Saint Paul, Minnesota
  - Columbia University Irving Medical Center - Herbert Irving Pavilion Site#104, New York, New York
  - University of Pennsylvania-Abramson Cancer Center Site#113, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center Site #102, Houston, Texas
  - NEXT Oncology Site #101, San Antonio, Texas
  - Virgnia Cancer Specialists Site #103, Fairfax, Virginia